CLINICAL TRIAL: NCT00945542
Title: Formula-driven vs Laboratory-guided Transfusion Practices in Bleeding Trauma Patients: A Feasibility Randomized Controlled Study
Brief Title: The Trauma- Formula-Driven Versus Lab-Guided Study (TRFL Study)
Acronym: TRFL
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: Canadian Department of National Defence (Other Government); Canadian Blood Services (Other); National Blood Foundation (Unknown)
Responsible Party: Principal Investigator, Dr. Jeannie Callum, Transfusion Medicine Specialist, Sunnybrook Health Sciences Centre
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 461-2008
Record Dates: First submitted 2009-07-22; First posted 2009-07-24 (Estimated); Last update posted 2011-12-02 (Estimated); Status verified 2011-12

CONDITIONS: Hemorrhagic Shock; Trauma Coagulopathy
Keywords: Trauma; Coagulopathy; Transfusion; Plasma; Massive Transfusion
MeSH Terms: conditions — Shock, Hemorrhagic; Wounds and Injuries; Hemostatic Disorders | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard of care (Other): Patients randomized to this arm will be treated as per Sunnybrook's current standard of care massive transfusion protocol. Crystalloid and red cell transfusions are performed to maintain volume status, and to maintain haemoglobin levels above 70 g/L. FFP is transfused based in 3-4 unit aliquots, for INR>1.5. Platelets are transfused 1 pool at a time (4 units Buffy coat platelets) to maintain platelet counts above 50 x 109/mL. Cryoprecipitate is transfused 8-12 units at a time to keep fibrinogen above 0.8 gram/L.
  Interventions: Other: Standard of care
- Preemptive transfusion (Experimental): Patients randomized to this arm will be transfused based on a pre-defined massive transfusion protocol. Blood bank will release blood a pre-defined packages. Blood will be received in aliquots containing 4 units off FFP, 1 pool of buffy coat platelet (4 units) and 4 units of RBC. This corresponds to an FFP:RBC transfusion ratio of 1:1.
  Patients randomized to the study protocol will be receiving the FFP and PTL at pre-defined ratios to RBC (1:1:1) up to 12h of hospitalization or earlier if cessation of the massive transfusion requested at the discretion of the treating physicians.
  Interventions: Other: Massive transfusion protocol

INTERVENTIONS:
Other: Massive transfusion protocol — Patients randomized to this arm will be transfused based on a pre-defined massive transfusion protocol. Blood bank will release blood a pre-defined packages. Blood will be received in aliquots containing 4 units off FFP, 1 pool of buffy coat platelet (4 units) and 4 units of RBC. As discussed previously, this would correspond to an FFP:RBC transfusion ratio of 1:1.
  Patients randomized to the study protocol will be receiving the FFP and PTL at pre-defined ratios to RBC (1:1:1) up to 12h of hospitalization or earlier if cessation of the massive transfusion requested at the discretion of the treating physicians.
  Other Names: Early and aggressive FFP transfusion; 1:1, FFP:RBC transfusion; Damage Control Resuscitation; Hemostatic Resuscitation; Early use of FFP
  Arms: Preemptive transfusion
Other: Standard of care — Patients randomized to this arm will be treated as per Sunnybrook's current standard of care massive transfusion protocol. Crystalloid and red cell transfusions are performed to maintain volume status, and to maintain haemoglobin levels above 70 g/L. FFP is transfused based in 3-4 unit aliquots, for INR>1.5. Platelets are transfused 1 pool at a time (4 units Buffy coat platelets) to maintain platelet counts above 50 x 109/mL. Cryoprecipitate is transfused 8-12 units at a time to keep fibrinogen above 0.8 gram/L.
  Arms: Standard of care

SUMMARY:
Background: Bleeding and coagulopathy still accounts for the majority of early in-hospital deaths following trauma. There have been lately several published studies suggesting that higher transfusion ratios of fresh frozen plasma (FFP), platelets (PTL) and cryoprecipitate (CRYO) to red blood cell (RBC) are associated with survival advantages. However, the evidence comes from retrospective data limited by a significant number of unaddressed confounders. In addition, the use of blood products bears known and important risks of complications.

Hypothesis: The adoption of a formula-driven transfusion practice with pre-defined ratios of FFP to PTL to RBC transfusion (1:1:1) is feasible and superior to current laboratory-guided transfusion practice in treating and/or preventing early coagulopathy improving survival rates in massively bleeding trauma patients .

Objective: To exam the feasibility of implementing a pre-defined ratio of FFP to PTL to RBC (1:1:1) transfusion protocol and its impact on a population of bleeding trauma patients.

Design: A two-year pilot feasibility randomized control trial at Sunnybrook Health Sciences Centre. Randomization: 70 patients are expected to be randomized to lab-driven or to formula-driven massive transfusion protocol and followed-up to 28 days or hospital discharge.

Study outcomes: protocol violation; in-hospital mortality by exsanguination; death at 28 days; coagulation competence defined by current standard coagulation tests (INR & PTT < 1.5 times normal; PTL ≥ 50 and Fibrinogen ≥ 1.0) or clotting factor levels ≥ 30%; correlation of current standard coagulation tests with clotting factors levels; cessation of bleeding; incidence of ALI, sepsis, MOF, transfusion-related circulatory overload, transfusion reactions; Ventilator-free days; ICU & Hospital LOS; thromboembolic events.

Intervention protocol: Transfusion of pre-defined ratios of FFP and PTL to RBC (1:1:1) (formula-driven) for the first 12h of hospitalization without coagulation tests guidance while patient is hemorrhaging or before if bleeding stops.

Statistical analysis: protocol compliance rate and in-hospital mortality rates within 24h and at 28 days will be assessed using Chi-square test. ROC analysis will be used to analyze coagulation competence.

Main expected outcomes: implementation of a formula-driven transfusion protocol is feasible and coagulation competence will be achieved faster and more efficiently in the study group.

ELIGIBILITY:
Inclusion Criteria

Patients were eligible for this study if they:

i) were adult trauma patients assessed by the trauma team; and ii) suffered either penetrating or blunt mechanism of injury; and

1. were bleeding and expected to require massive transfusion (either 4 units within the next 2 hours or ≥ 10 units of RBC in 24 h) or required transfusion of un-cross matched emergency stock red blood cells; and
2. had an episode of hypotension (systolic bp ≤ 90mmHg).

Exclusion Criteria

Patients were excluded if:

i) they were assessed in the trauma room more than six hours after injury; or ii) they received more than two units of RBC transfusion prior to arrival; or iii) they had suffered a concomitant severe brain injury (defined as any of the following: Glasgow Coma Scale of 3 due to severe traumatic brain injury; clear indication of immediate neurosurgical intervention based on clinical findings, mechanism of trauma associated with focal signs (anisocoria, CT evidence of intracranial bleeding with mass effect); or iv) they had evidence of having a catastrophic head injury (such as transcranial gunshot wound, open skull fracture with exposure/loss of brain tissue, or expert opinion by either the trauma team leader or neurosurgical consultant based on initial clinical or initial CT findings); or v) they had evidence that their shock state was unrelated to hemorrhage (ie cardiogenic, septic, anaphylactic, acute adrenal insufficiency, neurogenic, or obstructive (cardiac tamponade, tension pneumothorax and massive pulmonary emboli); or vi) they had a known hereditary or acquired coagulopathy unrelated to the trauma resuscitation (for example: hemophilia, hepatic insufficiency, or anti-coagulant medications); or vii) they were moribund with evidence of unsalvageable injuries.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2009-07; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Protocol compliance | 12 hours

SECONDARY OUTCOMES:
Mortality by Exsanguination; Hospital mortality; Cessation of Bleeding; Coagulation competence; Multiple Organ Dysfunction; Transfusion complications. | early and at 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Sandro B Rizoli, MD PhD, Principal Investigator — Sunnybrook Health Sciences Centre; Gordon D Rubenfeld, MD, MSc, Principal Investigator — Sunnybrook Health Sciences Centre; Homer C Tien, MD, MSc, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Nascimento B, Callum J, Tien H, Rubenfeld G, Pinto R, Lin Y, Rizoli S. Effect of a fixed-ratio (1:1:1) transfusion protocol versus laboratory-results-guided transfusion in patients with severe trauma: a randomized feasibility trial. CMAJ. 2013 Sep 3;185(12):E583-9. doi: 10.1503/cmaj.121986. Epub 2013 Jul 15. PMID 23857856
- [Derived] Nascimento B, Rizoli S, Rubenfeld G, Lin Y, Callum J, Tien HC. Design and preliminary results of a pilot randomized controlled trial on a 1:1:1 transfusion strategy: the trauma formula-driven versus laboratory-guided study. J Trauma. 2011 Nov;71(5 Suppl 1):S418-26. doi: 10.1097/TA.0b013e318232e591. PMID 22071998